CLINICAL TRIAL: NCT05743634
Title: A Phase I/II,Multicenter, Randomized, Double-Blind, Placebo and Active-Controlled Study to Evaluate the Safety,Efficacy and Immunogenicity of Recombinant Botulinum Toxin Type A for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: A Phase I/II Study of Recombinant Botulinum Toxin Type A for the Treatment of Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chongqing Claruvis Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YY001-001; CTR20221419 (Registry Identifier: www.chinadrugtrials.org.cn)
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Moderate to Severe Glabellar Lines
Keywords: YY001; Botulinum Toxin; Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Placebo and active controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group (Experimental): Single injection with YY001 in glabellar lines
  Interventions: Biological: YY001
- Active-Controlled Group (Active Comparator): Single injection with BOTOX® in glabellar lines
  Interventions: Biological: OnabotulinumtoxinA
- Placebo-Controlled Group (Placebo Comparator): Single injection with placebo in glabellar lines
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: YY001 — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Treatment Group
Biological: OnabotulinumtoxinA — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Active-Controlled Group
Biological: Placebo — Single treatment,intramuscularly injected into five sites.The total injection volume is 0.25 ml,0.05 ml per site.
  Arms: Placebo-Controlled Group

SUMMARY:
This is a phase 1/2, multicenter, randomized, double-blind, active-controlled and placebo-controlled study to evaluate safety,immunogenicity and efficacy of YY001 for the treatment of moderate to severe glabellar lines in male and female subjects of Chinese origin. The study has been designed to test the safety,efficacy,immunogenicity of YY001,and compare to onabotulinumtoxinA (BOTOX®) and placebo, in improving the appearance of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects from ≥18 to ≤65 years of age when signing an informed consent.
2. At screening and baseline,the subject has moderate to severe GL (grade of 2 or 3 on the 4-point Scale) at maximum frown when assessed by both the Investigator and the subject.
3. Agree to take part in the clinic trial and sign the informed consent form voluntarily.
4. Is able to observe the protocol by Investigator's assessment.
5. Male and female of childbearing potential agree to use a highly effective contraceptive method for the duration of the study(such as tubal ligation,abstinence,Intrauterine device,hormone,barrier method).For female of childbearing potential,her blood pregnancy test is negative within 7 days prior to study treatment,and urine pregnancy test is negative within 3 days prior to study treatment.Male can't donate the sperm within 3 months after treatment.

Exclusion Criteria:

1. Known allergy or hypersensitivity to any component of the study products(YY001 or BOTOX®).
2. Previous use of any cosmetic therapy in the glabella or forehead area,such as hyaluronic acid,phototherapy,hydrating needle,microneedle,chemical peeling,scar removal surgery or skin dermabrasion within 6 months before screening.Previous use of biodegradable filler within 12 months before screening,such as collagen,polylactic acid or calcium hydroxyapatite.Previous use of autologous fat, any permanent products (such as silicone, polyacrylamide,no matter how long the interval is) ,face-lift,or semi-permanent prosthesis.Planned use of any cosmetic therapy in the glabella or forehead area during the study(other than the study products).
3. Previous use of any botulinum toxin within 6 months prior to screening,or plan to use any botulinum toxin during the study(other than the study products).
4. Use of any non-steroid anti-inflammatory drug or anticoagulant within 1 week prior to study treatment.
5. Use of medications that affect neuromuscular transmission within 4 weeks prior to screening, such as muscle relaxant,aminoglycoside antibiotics,anticholinergic drugs,benzodiazepines,etc.
6. Probably use of prohibited drug during the study,as assessed by the investigator.
7. Abnormal skin at in the treatment area,scar or physical scars, in the investigator's opinion,may interfere with study evaluations.
8. Inability to substantially spread glabellar lines apart by surgery or finger smoothing, as determined by the investigator.
9. Ptosis,excessive facial asymmetry and skin laxity ,at screening and baseline.
10. History of facial nerve palsy.
11. Any medical condition that may interfere neuromuscular function including myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis, dysphagia,dyspnea,diplopia,angle-closure glaucoma,eyelid or eyebrow ptosis,etc.
12. Any concomitant disease including,unfit for the study by the investigator.
13. In acute attack.
14. Abnormal lab findings,and unfit for the study in the opinion of the investigator.
15. History of alcohol or drug abuse.
16. History of epilepsy.
17. Any severe psychiatric illness ,in the investigator's opinion, could affect the subject's participation in the study.
18. Female who is pregnant,or breast feeding.
19. In any other clinical study ,or Participated in any other interventional study within 30 days or 5 half-lives prior to screening.
20. Contract research organization,study site personnel or close relatives of the study site personnel , employees or close relatives of employees at the sponsor company.
21. Other conditions, in the Investigator's opinion, unfit for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Phase1:The incidence rate of adverse events and severe adverse events within 28 days after injection | Within 28 days
Phase1:The incidence rate of injection site reaction within 28 days after injection | Within 28 days
Phase1:The incidence rate of abnormal lab findings which have clinical significance within 28 days after injection | Within 28 days
Phase2:The response rate will be evaluated at 28 days by investigator at maximum frown | 28 days
  A response rate is defined as a subject who achieves a score of 0 or 1 in GL severity at maximum frown and at least 2 grades improvement from baseline by investigator's assessment
Phase2:The incidence rate of adverse events and severe adverse events within 12 weeks after injection | within 12 weeks
Phase2:The incidence rate of injection site reaction within 12 weeks after injection | within 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Qingfeng Li, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (6):
- China (6):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Nanfang Hospital,Southern Medical University, Guangzhou, Guangdong
  - Shanghai Ninth People's Hospital,Shanghai JiaoTong University school of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No